CLINICAL TRIAL: NCT00701090
Title: A Phase III, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of the Addition of Sitagliptin Compared With the Addition of Glimepiride in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin
Brief Title: A Study to Test the Safety and Efficacy of Sitagliptin Compared to Glimepiride in Patients With Type 2 Diabetes on a Stable Dose of Metformin (0431-803)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-803; 2008_503
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus, Non Insulin Dependent; Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 Diabetes Mellitus; Non Insulin Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): sitagliptin
  Interventions: Drug: sitagliptin; Drug: open-label metformin
- 2 (Active Comparator): glimepiride
  Interventions: Drug: Comparator: glimepiride; Drug: open-label metformin

INTERVENTIONS:
Drug: sitagliptin — Sitagliptin 100 mg q.d. (q.d. = once daily); Duration of Treatment: 30 weeks
  Other Names: Januvia
  Arms: 1
Drug: Comparator: glimepiride — glimepiride 1 mg per day to be up-titrated (up to week 18 of the double-blind treatment period) as considered appropriate by the investigator, based upon the results of patient's self blood glucose monitoring (SBGM). The maximum dose of glimepiride must not be higher than 6 mg/day.
  Arms: 2
Drug: open-label metformin — open-label metformin oral tablets (≥1500 mg/day) in addition to Glimepiride or Sitagliptin treatment.
  Other Names: metformin

SUMMARY:
A study to see if better control of type 2 diabetes can occur in patients taking a stable dose of metformin when they are also provided either sitagliptin or glimepiride. This study will also see if this treatment is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with type 2 diabetes
* On a stable dose of metformin of at least 1500 mg per day

Exclusion Criteria:

* History of type 1 diabetes
* Pregnant
* HIV positive
* On a weight loss program or medication
* Has a history of blood disorder, certain cancers, heart, liver or kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Arechavaleta R, Seck T, Chen Y, Krobot KJ, O'Neill EA, Duran L, Kaufman KD, Williams-Herman D, Goldstein BJ. Efficacy and safety of treatment with sitagliptin or glimepiride in patients with type 2 diabetes inadequately controlled on metformin monotherapy: a randomized, double-blind, non-inferiority trial. Diabetes Obes Metab. 2011 Feb;13(2):160-8. doi: 10.1111/j.1463-1326.2010.01334.x. PMID 21199268
- [Derived] Ommen ES, Xu L, O'Neill EA, Goldstein BJ, Kaufman KD, Engel SS. Comparison of treatment with sitagliptin or sulfonylurea in patients with type 2 diabetes mellitus and mild renal impairment: a post hoc analysis of clinical trials. Diabetes Ther. 2015 Mar;6(1):29-40. doi: 10.1007/s13300-015-0098-y. Epub 2015 Jan 30. PMID 25633134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 14-May-2008; Last Patient Last Visit: 27-Oct-2009; 109 study centers worldwide
Pre-assignment Details: Patients at least 18 years of age with type 2 diabetes mellitus with inadequate glycemic control (A1C ≥6.5 and ≤9.0%) on a stable dose of metformin (at a dose of at least 1500 mg per day for at least 12 weeks) were eligible to enter the 30 week study. Up to a 2 week screening period, followed by a 2-week placebo run-in.
Groups:
- Sitagliptin: The Sitagliptin 100 mg q.d. (q.d. = once daily) group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily (blinded) in addition to ongoing treatment with open-label metformin oral tablets (≥1500 mg/day).
- Glimepiride: The Glimepiride group includes data from patients randomized to receive treatment starting with 1 mg oral tablets of glimepiride (blinded) up-titrated until Week 18 as needed to a maximum dose of 6 mg q.d. in addition to ongoing treatment with open-label metformin oral tablets (≥1500 mg/day).
Period: Overall Study
Arm/Group | Sitagliptin | Glimepiride
Started | 516 | 519
Completed | 468 | 468
Not Completed | 48 | 51
Not completed — Adverse Event | 11 | 2
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 5 | 4
Not completed — Lost to Follow-up | 9 | 9
Not completed — Physician Decision | 3 | 4
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 11 | 16
Not completed — Other | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Glimepiride | Total
Number analyzed (Participants) | 516 | 519 | 1035
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.7) | 56.2 (10.1) | 56.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 240 | 472
  Male | 284 | 279 | 563
Race/Ethnicity, Customized [Number; unit: participants]
  White | 297 | 298 | 595
  Black | 6 | 6 | 12
  Asian | 109 | 111 | 220
  American Indian/Alaska Native | 25 | 26 | 51
  Other | 79 | 78 | 157
A1C (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 7.50 (0.70) | 7.51 (0.76) | 7.50 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 30
Description: Patient-level HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 30 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Week 0 to Week 30
Population: The per protocol population included all patients with a baseline value, a measurement at Week 30, and no major protocol violations (i.e., drug compliance <85%, use of prohibited medications, change of Metformin dose, incorrect double-blind study medication).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 443 | 436
Percent | -0.47 [-0.55 to -0.39] | -0.54 [-0.62 to -0.45]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Non-Inferiority or Equivalence — The pre-specified non-inferiority margin was 0.4%, i.e., Sitagliptin was declared non-inferior to glimepiride if the upper limit of the two-sided 95% confidence interval for the between group difference (sitagliptin minus glimepiride) was less than 0.4%; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.03 to 0.16], Standard Deviation 0.70 — ANCOVA model with terms: treatment, country, and baseline HbA1c

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 30
Description: Change from baseline at Week 30 was defined as Week 30 minus Week 0.
Time Frame: Week 0 to Week 30
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 446 | 444
mg/dL | -14.6 [-17.9 to -11.2] | -17.5 [-20.8 to -14.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; Mean Difference (Net) = 2.9, 95% CI 2-sided [-0.9 to 6.7], Standard Deviation 28.8 — ANCOVA model terms: treatment, country, and baseline

3. Secondary Outcome: Percent of Patients With at Least One Hypoglycemia Episode of Any Type at Week 30
Time Frame: Week 0 to Week 30
Population: All patients who took at least one dose of study therapy.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 516 | 518
Percentage of Participants | 7.0 | 22.0
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p < 0.001, Miettinen &Nurminen method; Risk Difference (RD) = -15.0, 95% CI 2-sided [-19.3 to -10.9] — Miettinen &Nurminen method was used for the 95% confidence interval

4. Secondary Outcome: Change From Baseline in Body Weight at Week 30
Description: Change from baseline at Week 30 was defined as Week 30 minus Week 0.
Time Frame: Week 0 to Week 30
Population: All patients who took at least one dose of study therapy and had body weight measurements at both baseline and Week 30.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 465 | 461
Kilograms | -0.8 [-1.1 to -0.5] | 1.2 [0.9 to 1.5]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, country, and baseline; Mean Difference (Net) = -2.0, 95% CI 2-sided [-2.3 to -1.6], Standard Deviation 2.9 — ANCOVA model terms: treatment, country, and baseline

5. Secondary Outcome: Percent of Patients With A1C <7.0% at Week 30
Time Frame: Week 30
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 443 | 436
Percentage of Participants | 52.4 | 59.6
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.47 to 0.90] — The parameter estimate and 95% CI represent the odds of having A1C <7.0% at Week 30 in the Sitagliptin group vs. the Glimepiride group, computed using a logistic regression model controlling for treatment, country and baseline A1C

6. Secondary Outcome: Percent of Patients With A1C <6.5% at Week 30
Time Frame: Week 30
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 443 | 436
Percentage of Participants | 21.2 | 27.5
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.47 to 0.95] — The parameter estimate and 95% CI represent the odds of having A1C <6.5% at Week 30 in the Sitagliptin group vs. the Glimepiride group, computed using a logistic regression model controlling for treatment, country and baseline A1C

ADVERSE EVENTS:
Description: Particpants analyzed are those who received at least 1 dose of study medication. One participant in the Glimepiride group did not receive any study medication and is not included in the analysis.
Arm/Group | Sitagliptin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 16/516 | 11/518
Other Adverse Events (participants affected / at risk) | 58/519 | 134/518
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=516) | Glimepiride (N=518)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Prostatitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=519) | Glimepiride (N=518)
Nasopharyngitis (Infections and infestations) | 25 | 36
Hypoglycaemia (Metabolism and nutrition disorders) | 36 | 114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.